CLINICAL TRIAL: NCT02912494
Title: A Phase III Study of JR-131 in Renal Anemia Patients With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Collaborators: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Masking: Double
Other Study IDs: JR-131-301
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- JR-131 (Experimental)
  Interventions: Drug: JR-131
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: JR-131
  Arms: JR-131
Drug: Darbepoetin alfa
  Arms: Darbepoetin alfa

SUMMARY:
The purpose of this study is to investigate the equivalence of JR-131 to Darbepoetin alfa and evaluate the safety of JR-131 in renal anemia patients with chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated with Darbepoetin alfa.

Exclusion Criteria:

* Patients having complication or history of a cardiovascular / lung / brain infarction.
* Patients having a pronounced hemorrhagic lesion.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Hemoglobin level | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280